CLINICAL TRIAL: NCT00002474
Title: Phase II Study of High Dose Cyclophosphamide, Mitoxantrone, and Carboplatin With Autologous Bone Marrow Transplantation in Refractory or Relapsed Ovarian Carcinoma
Brief Title: Combination Chemotherapy and Bone Marrow Transplant in Treating Patients With Refractory or Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: LUMC-3007; CDR0000076845 (Registry Identifier: PDQ (Physician Data Query)); NCI-V91-0058
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2003-03

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Cyclophosphamide; Mitoxantrone

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: mitoxantrone hydrochloride
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, carboplatin, and mitoxantrone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy with autologous bone marrow transplant may allow the doctor to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy and autologous bone marrow transplant work in treating patients with refractory or recurrent ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, duration of response, and overall survival of patients with refractory or relapsed ovarian epithelial cancer treated with high-dose cyclophosphamide, carboplatin, and mitoxantrone followed by autologous bone marrow transplantation.
* Determine the nonhematopoietic toxicity of this regimen in these patients.

OUTLINE: Autologous bone marrow is harvested before study entry. Patients receive high-dose cyclophosphamide IV over 1 hour and mitoxantrone IV over 15 minutes on days -8, -6, and -4 and carboplatin IV continuously on days -8 to -3 in the absence of unacceptable toxicity. Bone marrow is reinfused on day 0 beginning at least 60 hours after completion of carboplatin infusion.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 1.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of refractory or relapsed ovarian epithelial cancer

  * Must have failed prior regimen containing cisplatin or carboplatin
* Bidimensionally measurable or evaluable disease

  * Serial CA-125 antigen titers or cytologically positive pleural effusion and/or ascites acceptable as evaluable disease
* Autologous bone marrow harvest of greater than 1.2 x 10 to the eighth nucleated cells/kg required before study entry
* No evidence of tumor at marrow harvest sites by bilateral bone marrow aspirates and biopsies, pelvic x-ray, and bone scan
* CNS involvement allowed

PATIENT CHARACTERISTICS:

Age:

* Under 65

Performance status:

* SWOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* WBC greater than 3,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT and SGPT less than 2 times upper limit of normal

Renal:

* Creatinine clearance greater than 60 mL/min
* No prior hemorrhagic cystitis

Cardiovascular:

* LVEF greater than 45% by MUGA scan

Other:

* No hearing loss in voice tones
* No active infection
* No psychological contraindication to study treatment
* Not pregnant
* Negative pregnancy test
* HIV negative
* General medical condition must allow general anesthesia

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior bone marrow transplantation
* More than 4 weeks since other prior biologic therapy and recovered

Chemotherapy:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (at least 6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* More than 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Max Age: 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1991-02; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Response rate
Response duration
Overall survival
Nonhematopoietic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Stiff, MD, Study Chair — Loyola University
Locations (1):
- Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Result] Stiff PJ, Bayer R, Kerger C, Potkul RK, Malhotra D, Peace DJ, Smith D, Fisher SG. High-dose chemotherapy with autologous transplantation for persistent/relapsed ovarian cancer: a multivariate analysis of survival for 100 consecutively treated patients. J Clin Oncol. 1997 Apr;15(4):1309-17. doi: 10.1200/JCO.1997.15.4.1309. PMID 9193322
- [Result] Stiff P, Bayer R, Camarda M, Tan S, Dolan J, Potkul R, Loutfi S, Kinch L, Sosman J, Peace D, et al. A phase II trial of high-dose mitoxantrone, carboplatin, and cyclophosphamide with autologous bone marrow rescue for recurrent epithelial ovarian carcinoma: analysis of risk factors for clinical outcome. Gynecol Oncol. 1995 Jun;57(3):278-85. doi: 10.1006/gyno.1995.1143. PMID 7774830